CLINICAL TRIAL: NCT04928612
Title: An Open-Label, Non-randomized, Multi-center Phase I Study Evaluating the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Bi-Ligand-Drug Conjugate CBP-1018 in Patients With Advanced Solid Tumors
Brief Title: A Study of CBP-1018 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Coherent Biopharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBP-1018-101
Record Dates: First submitted 2021-05-29; First posted 2021-06-16 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part A -CBP-1018 Dose escalation/Part B- CBP-1018 monotherapy (Experimental): Part A: CBP-1018 administrated iv Q 2 W (4 weeks/cycle), utilizing accelerated titration at lower doses (0.03 mg/kg and 0.06 mg/kg) and an i 3+3 design at following doses (0.08 mg/kg,0.10 mg/kg,0.12 mg/kg and 0.14 mg/kg, etc.), respectively.
  Part B：Further evaluate the efficacy and safety profile of CBP-1018 in 4 tumor-specific cohorts.Cohort 1 (Metastatic castration resistant prostate cancer, mCRPC)；(Advanced renal cell cancer, RCC); Cohort 3 (Advanced lung cancer, LC); Cohort 4 (Other advanced solid tumors).
  Interventions: Drug: CBP-1018

INTERVENTIONS:
Drug: CBP-1018 — CBP-1018 for injection, IV infusion

SUMMARY:
This is an open-label, non-randomized, multi-center, phase I study of bi-ligand-drug conjugate CBP-1018 in patients with advanced solid tumors. This study will be conducted in 2 parts: Part A (Dose Escalation) and Part B (Dose Expansion). Both parts include screening period, treatment period, end of treatment (EOT)/withdrawal, safety follow-up (SFU) and long-term-follow-up (LTFU). CBP-1018 will be administrated on eligible subjects until disease progression, unacceptable toxicity, withdrawal of consent or Sponsor's decision to stop the study, etc.

DETAILED DESCRIPTION:
Part A (Dose Escalation) is to evaluate the safety, tolerability, PK and preliminary efficacy of CBP-1018 and determine the MTD and RP2D of CBP-1018 administrated iv Q2W (4 weeks/cycle), utilizing accelerated titration at lower doses (0.03 mg/kg and 0.06 mg/kg) and an i3+3 design at following doses (0.08 mg/kg,0.10 mg/kg,0.12 mg/kg and 0.14mg/kg, etc.), respectively. The DLT evaluation period will be 28 days from the first dose of CBP-1018. Up to 2 subjects will be allowed under DLT evaluation period at the same time. The interval between the first treatment of CBP-1018 to the 2 subjects under DLT evaluation period at the same time, is at least 1 week. Safety monitoring committee (SMC), comprised of Investigators and sponsor's medical personnel, etc., will be responsible for safety monitoring, dose escalation safety review and justification, MTD/RP2D determination, and other critical study decisions. A higher dose level may be added on the decision of SMC, if MTD is not observed at 0.14mg/kg. Intermediate dose levels among planned dose levels may also be added by SMC for further exploration. RP2D may be the same dose level as MTD or lower than it. Up to 10 additional subjects will be enrolled in one or more dose levels that have been shown to be safe and tolerable to better estimate the RP2D and better characterize the safety, efficacy, and pharmacodynamics for CBP-1018. Different schedules (QW or Q3W, for example) may be explored in Part A, according to emerging clinical and PK data, either.

Part B (Dose Expansion) is to further evaluate the efficacy and safety profile of CBP-1018 in 4 tumor-specific cohorts:

• Cohort 1 (Metastatic castration resistant prostate cancer, mCRPC)；Cohort 2(Advanced renal cell cancer, RCC); Cohort 3 (Advanced lung cancer, LC); Cohort 4 (Other advanced solid tumors).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent (ICF) prior to any study-specific procedures.
* Men or women ≥ 18 years old when signed ICF.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Life expectancy of ≥ 3 months, in the opinion of the Investigator.
* Pathologically documented, advanced solid tumor including metastatic castration resistant prostate cancer (mCRPC), advanced renal cell cancer (RCC), advanced lung squamous cell cancer (LSCC), etc.
* Subjects must have received prior standard therapy appropriate for their tumor type and stage of disease, or in the opinion of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy.
* At least one non-irradiated measurable lesion per RECIST 1.1 or bone lesion per PCWG3 (only for mCRPC), optional for low dose level (≤ 0.08 mg/kg) of Part A.
* Available archived or fresh tumor tissue samples, optional for low dose level (≤ 0.08 mg/kg) of Part A.
* Adequate bone marrow and organ function, defined as:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, not requiring growth factor support for at least 28 days prior to the first dose of CBP-1018.
* Hemoglobin (Hb) ≥ 100 g/L, not requiring transfusion support for at least 14 days or growth factor support for at least 28 days prior to the first dose of CBP-1018.
* Platelet count ≥ 100 × 109/L, not requiring transfusion support for at least 7 days prior to the first dose of CBP-1018.
* Total bilirubin (TBIL) ≤ 1.5 × ULN, alkaline phosphatase (ALP) ≤ 1.5 × ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0× ULN if no demonstrable liver metastases.
* TBIL≤ 1.5 × ULN, ALT and AST ≤ 5.0 × ULN in the presence of liver metastases.
* TBIL < 2.0 × ULN for subjects with documented Gilbert's syndrome or < 3.0 × ULN for subjects for whom the indirect bilirubin level suggests an extrahepatic source of elevation.
* Creatinine ≤ 1.0 × ULN, or creatinine clearance ≥ 50 mL/min as calculated using Cockcroft-Gault formula.
* International Normalized Ratio (INR) ≤ 1.5 × ULN (within the therapeutic range for subjects receiving anticoagulation therapeutic) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
* LVEF ≥ 50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA).
* Female subjects of childbearing/reproductive potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of CBP-1018. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Male subjects of fathering potential and subjects of childbearing/reproductive potential must agree to use highly effective methods of contraception (see Appendix 4) throughout the study and for at least 30 days after the last dose of CBP-1018.

Exclusion Criteria:

* Known prior or suspected hypersensitivity to study drugs or any component in their formulations.
* Concurrent malignancy within 5 years prior to the first dose of CBP-1018, other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer not requiring treatment, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma.
* Active central nervous system (CNS) metastases. Previously diagnosed CNS metastases are eligible if have been treated and recovered from the acute effects of radiation therapy or surgery prior to the first dose of CBP-1018, have discontinued corticosteroid treatment for CNS metastases for at least 4 weeks and are neurologically stable.
* Major surgery, systemic anticancer therapy (chemotherapy, targeted therapy, immunotherapy, endocrine therapy, biotherapy) or participation in other therapeutic studies within 4 weeks prior to the first dose of CBP-1018.
* Radiotherapy administrated within 21 days prior to the first dose of CBP-1018, or localized palliative radiotherapy administered within 7 days prior to the first dose of CBP-1018.
* Any toxicities attributed to prior anti-cancer therapy, other than alopecia and fatigue, that have not resolved to Grade 1 (NCI CTCAE 5.0) or baseline prior to the first dose of CBP-1018.
* Poorly controlled concurrent diseases as diabetes, hypertension (systolic blood pressure >160 mmHg or diastolic blood pressure > 100 mmHg), etc.
* History of any of the following cardiovascular conditions within 12 months of enrollment: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association.
* History of clinically significant lung diseases as interstitial pneumonia, pneumonitis, pulmonary fibrosis, and severe radiation pneumonitis, or suspected to have these diseases by imaging at screening period.
* Active bleeding disorder or other history of grade ≥ 3 hemorrhage within 4 weeks prior to the first dose of CBP-1018.
* Requirement of anticoagulant therapy with oral vitamin K antagonists. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed. Therapeutic use of low molecular weight heparin is allowed.
* History of deep vein thrombosis or pulmonary embolism within 6 months prior to the first dose of CBP-1018.
* Active infection requiring intravenous (IV) antibiotics within 1 weeks prior to the first dose of CBP-1018.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Positive Hepatitis B Surface Antigen (HepBsAg) (indicative of chronic Hepatitis B), positive Hepatitis total core antibody with negative HepBsAg (suggestive of occult hepatitis B) or detectable Hepatitis C virus Ribonucleic acid (RNA) by PCR (Hepatitis C Antibody test for screening, followed by PCR for Hepatitis C virus RNA if HepCAb is positive).
* Live-virus vaccination within 30 days prior to the first dose of CBP-1018. Seasonal influenza vaccines that do not contain live virus are allowed.
* Current or anticipated need for treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers.
* History or current evidence of any other condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) in Part A | 12 months
  Incidence of dose limiting toxicity (DLTs), treatment-emergent adverse events (TEAE), treatment-related adverse events, serious adverse events (SAEs) and clinically significant changes in vital signs, physical examinations, electrocardiogram (ECGs), and clinical laboratory tests per the National Cancer Institute's Common Terminology Criteria for Adverse Events, version 5.0 (NCI CTCAE 5.0).
MTD of CBP-1018 in Part A | 12 months
  maximum tolerated dose（MTD）
Recommended Phase 2 dose (RP2D) of CBP-1018 in Part A | 12 months
  The recommended Phase 2 dose (RP2D) is defined as the dose level chosen by the sponsor (in consultation with the investigators) based on safety,tolerability, efficacy, PK data collected during the dose escalation study of CBP-1018.
ORR in Part B | enrollment to end of treatment up to 3 years
  ORR（Objective response rate） per RECIST 1.1 ,PCWG3 (only for bone lesions of prostate cancer)

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | 12 months
  Maximum serum concentration (Cmax) of CBP-1018 will be investigated.
Time to maximum serum concentration (Tmax) of CBP-1018 | 12 months
  Tmax of CBP-1018 will be investigated.
Elimination half-life (T1/2) of CBP-1018 | 12 months
  T1/2 of CBP-1018 will be investigated.
AUC0-t of CBP-1018 | 12 months
  AUC0-t is defined as area under the serum concentration-time curve from time 0 to the time of the last measurable concentration
Clearance (CL) in the serum of CBP-1018 per unit of time | 12 months
  CL in the serum of CBP-1018 per unit of time will be investigated
ORR in Part A | 12 months
  ORR（Objective response rate） per RECIST 1.1,PCWG3 (only for bone lesions of prostate cancer)
Immunogenicity assessment | enrollment to end of treatment up to 3 years
  Anti-drug antibody(ADA) against CBP-1018 will be evaluated.
Duration of Response (DOR) | enrollment to end of treatment up to 3 years
  The DOR is evaluated by investigator according to RECIST 1.1.,PCWG3 (only for bone lesions of prostate cancer).
Progression-free survival rate (PFS) | enrollment to end of treatment up to 3 years
  The PFS is evaluated by investigator according to RECIST 1.1.,PCWG3 (only for bone lesions of prostate cancer).
Disease Control Rate(DCR) | enrollment to end of treatment up to 3 years
  The DCR is evaluated by investigator according to RECIST 1.1.,PCWG3 (only for bone lesions of prostate cancer).

OTHER OUTCOMES:
Neuroendocrine or small cell transformation-associated markers of mCRPC | 12 months
  Neuroendocrine or small cell transformation-associated markers of mCRPC
Potential metabolites of CBP-1018 | 12 months
  Potential metabolites of CBP-1018 in human plasma, urine, feces, if appropriate.
Biomarkers | 12 months
  Biomarkers in tumor tissues with relationships of CBP-1018 efficacy/safety including,but not limited to, FOLR1
Biomarkers | 12 months
  Biomarkers in tumor tissues with relationships of CBP-1018 efficacy/safety including,but not limited to,PSMA

CONTACTS AND LOCATIONS:
Overall Officials: Hai Huang, Ph D, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Sun Yat-Sen memorial hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No